CLINICAL TRIAL: NCT00727987
Title: A Study of Golimumab (CNTO 148) Administered in Combination With Methotrexate (MTX) in Patients With Active Rheumatoid Arthritis
Brief Title: A Safety and Efficacy Study of Golimumab (CNTO 148) in Patients With Active Rheumatoid Arthritis Despite Methotrexate Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Collaborators: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR015340; JNS012-JPN-03 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Fully Human anti-TNFa monoclonal antibody; CNTO148; Golimumab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — golimumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CNTO 148 50 mg + methotrexate (Experimental)
  Interventions: Drug: CNTO 148; Drug: Methotrexate (MTX)
- CNTO 148 100 mg + methotrexate (Experimental)
  Interventions: Drug: Methotrexate (MTX)
- Placebo + methotrexate (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Methotrexate (MTX)

INTERVENTIONS:
Drug: CNTO 148 — 50 mg or 100 mg given as a subcutaneous (under the skin) injection once every 4 weeks up to Week 152.
  Other Names: Golimumab
  Arms: CNTO 148 50 mg + methotrexate
Drug: Placebo — Placebo identical in appearance to CNTO 148 given as a subcutaneous (under the skin) injection once every 4 weeks up to Week 24.
  Arms: Placebo + methotrexate
Drug: Methotrexate (MTX) — 6 mg/week to 8 mg/week taken orally (by mouth) from at least 4 weeks before the initial investigational treatment to the completion of assessment at Week 52.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of golimumab in patients with active rheumatoid arthritis despite Methotrexate therapy. Another objective is to evaluate the pharmacokinetics of golimumab.

DETAILED DESCRIPTION:
This clinical study is scheduled to be performed for the purpose of evaluating the safety and effectiveness of golimumab (CNTO148) administered in combination with stable dose (6-8mg/week) of methotrexate (MTX) to patients with rheumatoid arthritis (RA). CNTO148 50 mg group: CNTO148 50 mg SC injections every 4 weeks from the first administration until week 152. If early escape, 100 mg SC injections every 4 weeks from week 16 until week 152. CNTO148 100 mg group: CNTO148 100 mg SC injections every 4 weeks from the first administration until week 152 whether early escape or not Placebo group: Placebo SC injections every 4 weeks from the first administration until week 20 and then CNTO148 50mg SC injections every 4 weeks from week 16 until week 152

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with rheumatoid arthritis at least 3 months prior to registration and who are definitely identified as having rheumatoid arthritis, at the time of informed consent, according to the criteria for classification established by the American College of Rheumatology (1987)
* Patients in whom MTX therapy (>= 6 mg/week) was started more than 3 months before the first administration and who have been treated with MTX at a stable dose (6-8 mg/week) for at least 4 weeks before the first administration
* Patients having at least 4 swollen joints and at least 4 tender joints at the time of registration and immediately before the first administration.

Exclusion Criteria:

* Patients with a history of hypersensitivity to human immunoglobulin proteins or other ingredients of golimumab
* Patients who have previously experienced or are suffering from any of the following diseases: (i) Collagen diseases other than rheumatoid arthritis, (ii) Latent or active granulomatous infections such as histoplasmosis and coccidioidomycosis, (iii) Felty syndrome, etc
* Patients with a severe, advanced, or poorly controlled disease in any of the kidney, liver, blood, gastrointestinal system, endocrine system, lung, heart, nervous system, psychiatric system, and brain.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2008-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
ACR 20% response | Week 14

SECONDARY OUTCOMES:
ACR 50% response, ACR 70% response, ACR 90% response, Changes from the pretreatment values in the DAS (Disease Activity Score) 28, and the HAQ (Health assessment questionnaire) | Week 14

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (65):
- Japan (65):
  - Asahi
  - Asahikawa
  - Azumino
  - Chiba
  - Fukui
  - Fukuoka
  - Fukushima
  - Gifu
  - Goshogawara
  - Hachiōji
  - Hamamatsu
  - Higashi-Hiroshima
  - Hiki
  - Hiroshima
  - Hitachi
  - Iruma
  - Izumisano
  - Izumo
  - Kamakura
  - Katō
  - Kawachi-Nagano
  - Kawagoe
  - Kawasaki
  - Kita-Gun
  - Kitakyushu
  - Kitamoto
  - Kobe
  - Kumamoto
  - Kyoto
  - Matsue
  - Matsumoto
  - Matsuyama
  - Nagano
  - Nagasaki
  - Nagoya
  - Narashino
  - Nishinomiya
  - Ohta-Ku
  - Osaka
  - Ōita
  - Ōsaki
  - Sagamihara
  - Saitama
  - Sapporo
  - Sasebo
  - Sendai
  - Shimotsuga
  - Shimotsuke
  - Shinjuku
  - Shinjuku-Ku
  - Shizuoka
  - Suita
  - Tokorozawa
  - Tokushima
  - Tokyo
  - Toshima-Ku
  - Toyama
  - Toyoake
  - Toyohashi
  - Tsu
  - Tsukuba
  - Tsukubo
  - Ube
  - Yokohama
  - Yufu

REFERENCES:
- [Derived] Tanaka Y, Harigai M, Takeuchi T, Yamanaka H, Ishiguro N, Yamamoto K, Miyasaka N, Koike T, Kanazawa M, Oba T, Yoshinari T, Baker D; GO-FORTH Study Group. Golimumab in combination with methotrexate in Japanese patients with active rheumatoid arthritis: results of the GO-FORTH study. Ann Rheum Dis. 2012 Jun;71(6):817-24. doi: 10.1136/ard.2011.200317. Epub 2011 Nov 25. PMID 22121129
- See also: A Study of Golimumab (CNTO 148) Administered in Combination with Methotrexate (MTX) in Patients with Active Rheumatoid Arthritis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=426&filename=CR015340_CSR.pdf